CLINICAL TRIAL: NCT04583098
Title: The Effect of Fecal Microbiota Transplantation on the Decolonization of Carbapenem-resistant Enterobacteriaceae or Vancomycin-resistant Enterococci in the Gut
Brief Title: The Effect of Fecal Microbiota Transplantation on the Decolonization of Multidrug-resistant Organisms
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Seung Soon Lee, Associate Professor, Chuncheon Sacred Heart Hospital
Other Study IDs: 2020-08-006
Record Dates: First submitted 2020-09-27; First posted 2020-10-12 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection; Vancomycin-Resistant Enterococcal Infection
Keywords: Fecal Microbiota Transplantation; Carbapenem-Resistant Enterobacteriaceae; Vancomycin-Resistant Enterococci; Gastrointestinal Microbiome
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool (gut microbiota)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- carbapenem-resistant Enterobacteriaceae: FMT using frozen or capsulized stool
  Interventions: Other: fecal microbiota transplantation
- vancomycin-resistant Enterococci: FMT using frozen or capsulized stool
  Interventions: Other: fecal microbiota transplantation

INTERVENTIONS:
Other: fecal microbiota transplantation — frozen or capsulized stool from donors who had already finished recommended blood & stool screening for stool donors

SUMMARY:
The purpose of this study is to assess the effect of fecal microbiota transplantation for the decolonization of carbapenem-resistant Enterobacteriaceae or vancomycin-resistant Enterococci in the gut.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study exploring the decolonization effect of Fecal Microbiota Transplantation (FMT) in patients colonized with Carbapenem-resistant Enterobacteriaceae (CRE) and Vancomycin-resistant Enterococci (VRE).

Patients who have provided written consent for participation in the study will be required to maintain fasting starting from the evening before the procedure, after discontinuing broad-spectrum antibiotics for a minimum of 3-7 days. Subsequently, a bowel preparation will be carried out twice - the evening before and the morning of the procedure. Once the bowel preparation is complete, 1 hour before the procedure, patients will receive loperamide to reduce bowel movements and then proceed to the endoscopy suite.

Fecal microbiota transplantation (FMT) will be carried out with the acquired frozen donor stool, which will be thawed for 2 hours at room temperature following purchase and delivery from a stool bank, under the consent and supervision of the patient or guardian. Frozen stool from carefully screened donors who have passed the rigorous screening of both Stage 1 clinical assessment and Stage 2 laboratory tests (including evaluation for antibiotic resistance organisms) will be supplied from a stool bank of Microbiotix inc. (Hyun Soo Seo, et al. Ann Lab Med 2021;41:424-428).

The FMT procedure will be conducted in collaboration with the research team in the Division of Gastroenterology. During the procedure, no tissue biopsy or excessive endoscope insertion will be performed. The FMT involves the simple infusion of thawed donor stool into the terminal ileum under colonoscopy, which takes approximately 5-10 minutes. The procedure carries minimal risk of bleeding, perforation, or aspiration. In most cases, it will be performed under sedation with colonoscopy. If smooth insertion of the colonoscope or proper visualization of the colon is hindered, or if colonic preparation is not successful, Esophagogastroduodenoscopy (EGD) will be performed with sedation, and thawed donor stool will be infused into the third portion of the duodenum. This procedure also poses minimal risk of regurgitation or aspiration due to its anatomical and physiological characteristics. After the procedure, the lower extremities will be elevated by about 30 degrees to prevent the transplanted stool from exiting. A one-day fasting period will be maintained after the procedure to facilitate successful engraftment of the transplanted stool, followed by the gradual resumption of a regular diet. Following FMT, repeated rectal swab cultures will be conducted to confirm three consecutive negative results for CP-CRE or VRE at 3-7 day intervals.

In cases where encapsulated fecal material is used for FMT, it will be ingested along with high-acid cranberry or orange juice. The capsules are specially designed to dissolve in low-acidic environments, allowing them to reach the terminal ileum for safe administration without the need for bowel preparation. On the first day, 15 capsules will be consumed, followed by another 15 capsules on the second day, for a total of 30 capsules. Subsequently, repeated rectal swab tests will be conducted to confirm three consecutive negative results for CP-CRE or VRE at 3-day intervals.

According to patient random allocation, fecal samples and clinical metadata will be periodically collected (prior to FMT, 1 month, 3 months, 6 months, and 12 months after FMT) from both recipients and donors. These collected samples will undergo full-length 16S rRNA sequencing and shotgun metagenomic sequencing to comprehensively analyze the gut microbiome. Through this analysis, the aim is to elucidate the intestinal microorganisms associated with decolonization outcomes and mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 years-old with carbapenem-resistant Enterobacteriaceae(CRE) or vancomycin-resistant Enterococci(VRE) rectal colonization
* Patients who have received written informed consent for fecal microbiota transplantation and collection of stool samples

Exclusion Criteria:

* Patients who have not completed acute-phase treatment, including antibiotic treatment
* If patients are pregnant, may be pregnant, or are lactating
* Patients who have not received written informed consent for the study enrollment
* Patients who are judged to be unhelpful to participate in the study according to the researcher's judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CRE- or VRE-rectal colonizer who have given written informed consent for fecal microbiota transplantation and collection of stool samples for CRE or VRE decolonization
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
successful decolonization of carbapenem-resistant Enterobacteriaceae or vancomycin-resistant Enterococci in the gut within 3 months after fecal microbiota transplantation | within 3 months
  Successful decolonization of carbapenem-resistant Enterobacteriaceae or vancomycin-resistant Enterococci was defined as three consecutive, carbapenem-resistant Enterobacteriaceae or vancomycin-resistant Enterococci-negative surveillance rectal swab cultures repeated with a 3-day interval within 3 months after fecal microbiota transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Seung Soon Lee, MD, Principal Investigator — Chuncheon Sacred Heart Hospital
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided